CLINICAL TRIAL: NCT05462977
Title: Efficacy of Rhythmically Entrained Exercise in Community-Dwelling Older Adults
Brief Title: Rhythmically Entrained Exercise in Community-Dwelling Older Adults
Acronym: REECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FY22-106
Record Dates: First submitted 2021-10-13; First posted 2022-07-18 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Exercise; Gait; Cognitive Decline; Caregiver Burden; Cognitive Impairment; Dementia; Alzheimer Disease; Mild Cognitive Impairment; Respite Care; Mental Health; Depression; Music Therapy; Psychosocial Intervention; Cognition; Geriatric Assessment; Cognitive Dysfunction; Cognitive Aging; Outcome Assessment, Health Care; Balance; Fall; Walking; Affect; Physical Exertion; Memory Deficit; Memory Disorders; Memory Impairment; Neuropsychological Tests; Executive Function; Middle Aged; Healthy Aging; Elderly
Keywords: Physical Activity; Rhythmic Entrainment; Synchronous Music; Rhythmic Auditory Stimulation; Rhythmic Auditory Cue; Gait Training; Mobility; Movement; Perceived Exertion; Musical Pleasure; Groove; Memory; Executive Function; Older Adults
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction; Caregiver Burden; Dementia; Alzheimer Disease; Psychological Well-Being; Depression; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be invited to participate in a music-based group exercise program for 20 weeks (30 - 40 min/day, up to 6 days/week).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group exercise with beat-accented synchronous music stimulation (Experimental): Participants will be asked to participate in a music-based group exercise program for 24 weeks (up to 6 days/week, 30 - 45 min/day), which is designed for older adults with functional limitations to safely exercise on a chair or in a supported standing posture for the improvement of aerobic capacity, upper and lower body strength, and balance control at a gradually increasing pace based on the tempo of the beat-accented synchronous music playlists.
  Interventions: Behavioral: Group exercise program

INTERVENTIONS:
Behavioral: Group exercise program — Participants will be asked to join a music-based group exercise program for 24 weeks (up to 6 days/week, 30 - 45 min/day), which is designed for older adults with functional limitations to safely exercise on a chair or in a supported standing posture for the improvement of aerobic capacity, upper and lower body strength, and balance control at a gradually increasing pace in synchrony with music.

SUMMARY:
Researchers at the University of North Carolina at Greensboro conduct a single-arm intervention trial to investigate the efficacy of a music-based group exercise program for community-dwelling older adults. Up to forty participants will be recruited to participate in a music-based light-to-moderate intensity group exercise program for 20 weeks (30 - 40 min/day, up to 6 days/week), which is designed for older adults with or without functional limitations to exercise with chairs for the improvement of aerobic capacity, upper and lower body strength, and balance control at a gradually increasing pace. During the exercise sessions, participants will be trained to move in time with music playlists in synchronous tempos. Primary outcomes are cognitive performance, mobility, and health-related quality of life measured before and after the intervention. Secondary outcomes are adherence to the exercise program as a potential mediator of the treatment.

DETAILED DESCRIPTION:
Researchers at the University of North Carolina at Greensboro are conducting a single-arm intervention trial to investigate the efficacy of a music-based group exercise program for community-dwelling older adults. Up to forty participants will be recruited to participate in a music-based light-to-moderate intensity group exercise program for 20 weeks (30 - 40 min/day, up to 6 days/week), which is designed for older adults with or without functional limitations to exercise with chairs for the improvement of aerobic capacity, upper and lower body strength, and balance control at a gradually increasing pace. During the exercise sessions, participants will be trained to move in time with music playlists in synchronous tempos. Primary outcomes are cognitive performance, mobility, and health-related quality of life measured before and after the intervention. Secondary outcomes are adherence to the exercise program as a potential mediator of the treatment. The research team aims to determine whether (1) a music-based light-to-moderate intensity group exercise intervention beneficially impacts mobility, cognitive function, and health-related quality of life in community-dwelling older adults; (2) the treatment effect is mediated by adherence to physical activity; and (3) the treatment effect is moderated by cognitive impairment or functional limitations.

ELIGIBILITY:
Inclusion Criteria:

* 55 - 99 years old
* Capable of being ambulatory with or without an assistive device.
* No cardiac or pulmonary conditions or any neurological or musculoskeletal comorbidity or pain that would make light-intensity exercise dangerous, determined by the Physical Activity Readiness Questionnaire for Everyone or confirmed by their local medical practitioner if necessary.
* Having adequate hearing for a conversation (including with hearing aids)
* Capable of following the study procedures
* No severe anxiety or depression
* Mild to moderate cognitive impairment

Exclusion Criteria:

* Age younger than 55 or older than 99
* Severe anxiety or depression
* Severe cognitive impairment

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of fall risks | Baseline and change from baseline at month 5
  Participants' fall risks will be measured by Timed Up & Go Test
Change of walking endurance | Baseline and change from baseline at month 5
  Participants' gait and walking endurance will be measured by 6-Minute Walk Test
Change of balance control | Baseline and change from baseline at month 5
  Participants' balance control will be measured by 4-Stage Balance Test
Change of lower body strength | Baseline and change from baseline at month 5
  Participants' lower body strength will be measured by 30-second Chair Stand Test
Change of cognitive function | Baseline and change from baseline at month 5
  Participants' cognitive function will be measured through Montreal Cognitive Assessment , Flanker Inhibitory Control and Attention test, and Pattern Comparison Processing Speed Test.
Change of health-related quality of life | Baseline and change from baseline at month 5
  EuroQol Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shin Park, PhD, Principal Investigator — University of North Carolina, Greensboro
Locations (1):
- UNC Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We don't have a plan to share IPD with other researchers at the moment.

REFERENCES:
- [Result] Park KS, Buseth L, Hong J, Etnier JL. Music-based multicomponent exercise training for community-dwelling older adults with mild-to-moderate cognitive decline: a feasibility study. Front Med (Lausanne). 2023 Aug 21;10:1224728. doi: 10.3389/fmed.2023.1224728. eCollection 2023. PMID 37671396
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fmed.2023.1224728/full